CLINICAL TRIAL: NCT05944107
Title: Impact on Anticoagulation Management When Activated Clotting Time is Combined With Heparin Concentration Monitoring in Cardiac Surgery: a Randomised Clinical Trial
Brief Title: Anticoagulation Management in Complex Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Anna Gkiouliava, Principal Investigator, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 3432
Record Dates: First submitted 2023-06-24; First posted 2023-07-13 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Extracorporeal Circulation
Keywords: anticoagulation; cardiopulmonary bypass; heparin; titration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activated Clotting Time (ACT) (Active Comparator): In this group, only ACT measurements and fixed doses of heparin and protamine are administered.
  ACT is measured using the ACT Plus device (Medtronic, MN, USA). Heparin formulation administered is HEPARIN/LEO INJ.SOL 25000IU/5ML. Protamine formulation administered is PROTAMINE SULPHATE/LEO PHARMA 10mg/ml
  Interventions: Other: Activated Clotting Time
- Heparin Concentration (HC) (Active Comparator): In this group, the Hepcon HMS Plus (Medtronic, MN, USA) is used to perform heparin concentration calculations and test each patient's individual response to heparin. Specifically tests performed were:
  * Heparin Dose Response test
  * Heparin Assay test
  Interventions: Other: Activated Clotting Time measurements combined with heparin concentration monitoring

INTERVENTIONS:
Other: Activated Clotting Time measurements combined with heparin concentration monitoring — In the HC group, the initial heparin dose is calculated using the HepCon HMS Plus . Except for ACT, heparin concentration is measured to maintain target heparin levels during CPB. The protamine dose for reversal is computed based on actual measured heparin levels using the device. ACT is also performed in all instances.
  Arms: Heparin Concentration (HC)
Other: Activated Clotting Time — The target ACT for procedures other than Coronary Artery Bypass Grafting (CABG) is 400s when Minimally Invasive Extracorporeal Circulation is used. A bolus of 300 International Units(IU)/kg heparin are administered to reach this target and initiate cardiopulmonary bypass (CPB). Repeated ACT measurements guide further heparin dose to maintain adequate anticoagulation. Then, at the end of the CPB, 0.75 mg of protamine are administered for every 100IU of the initial heparin bolus.
  Arms: Activated Clotting Time (ACT)

SUMMARY:
The goal of this clinical trial is to compare the anticoagulation management with or without heparin concentration level guidance, in patients undergoing valve or complex cardiac surgery during cardiopulmonary bypass using closed, coated circuits. The main questions it aims to answer are:

* initial heparin bolus, subsequent supplementary doses and total heparin variance among groups.
* protamine dose among groups.

Participants are adult patients scheduled for valve or complex cardiac surgery. They are randomised to either Activated Clotting Time guided management alone or combined with heparin level concentration monitoring.

ELIGIBILITY:
Inclusion Criteria:

* elective procedures
* cardiac surgery, except for Coronary Artery Bypass Grafting
* Cardiopulmonary bypass under Minimally Invasive Extracorporeal Circulation

Exclusion Criteria:

* known allergy to heparin or protamine
* hematological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Heparin dose | Bolus dose before cardiopulmonary bypass
  Heparin dose, IU
Heparin dose | Total dose after cardiopulmonary bypass
  Heparin dose, IU
Protamine dose | Total dose after cardiopulmonary bypass
  Protamine dose, mg

SECONDARY OUTCOMES:
Platelet count | Immediately after surgery
  Platelet count per mm^3
Platelet count | 24 hours after surgery
  Platelet count per mm^3
Platelet count | 48 hours after surgery
  Platelet count per mm^3

CONTACTS AND LOCATIONS:
Overall Officials: Helena Argiriadou, Dr, Study Director — AHEPA University Hospital, Aristotole University of Thessaloniki
Locations (1):
- AHEPA University Hospital, Aristotle University of Thessaloniki, Thessaloniki, Greece